CLINICAL TRIAL: NCT03424200
Title: Coaching for Cognition in Alzheimer's (COCOA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Institute for Systems Biology (Other); Arivale (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COCOA
Record Dates: First submitted 2018-01-10; First posted 2018-02-06 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching plus Routine Care (Other): Participants will receive coaching plus routine care
  Interventions: Other: Coaching plus routine care
- Routine Care (Other): Participants will receive the routine care
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Routine care — Participants will receive routine care
  Arms: Routine Care
Other: Coaching plus routine care — Participants will receive coaching plus routine care
  Arms: Coaching plus Routine Care

SUMMARY:
One major study objective is, using 2 study arms (data-driven health coaching plus RC vs. RC only), to evaluate the efficacy of data-driven health coaching. 'RC only' will serve as the control group. Participants will be enrolled in the trial on the basis of an existence of objective cognitive impairment defined by the MCI Screen (MCIS) and being in one of three functional stages as defined by the Functional Assessment Staging Test (FAST). The three FAST stages correspond to cognitive impairment without functional impairment (FAST 2), cognitive impairment with functional impairment without impairment in instrumental activities of daily living (FAST 3, also known as mild cognitive impairment, MCI), or cognitive impairment with impaired instrumental activities of daily living (FAST 4). Study objectives include measuring treatment related changes in cognitive and functional abilities, quality of life, and biological or biochemical measures.

A second major study objective is to analyze longitudinal multi-omic data from individuals on a trajectory of early-stage dementia, to discover correlations between measured variables, and identify models of causation that can further advance knowledge and research in brain degeneration and healthy living

DETAILED DESCRIPTION:
Up to 200 FAST Stages 2-4 patients with cognitive impairment will be randomized into data-driven health coaching vs. control groups. The participants will be treated and monitored for 24 months.

Subject Identification and Recruitment Study participants will be recruited from a high-volume memory clinic and a large physician medical group. Up to 200 participants will be enrolled in this prospective randomized study (up to 100 in each treatment arm).

Procedures for Obtaining Informed Consent All participants will receive the Experimental Research Subject's Bill of Rights prior to signing the informed consent form (ICF), authorization of use and disclosure of protected health information (PHI), and authorization of medical record release for the subject's treating physician, will be obtained from each participants prior to enrolling in the study. A copy of all signed ICF's will be given to the participants, and the investigator will retain the original.

FAST staging (see Attachment II for the FAST administrating and scoring) will be done before participants are consented to determine whether they or a legally appointed representative (LAR) can consent to participate in the study. In this study, participants with FAST stages 2-4 will be recruited (see Inclusion Criteria).

* Considerations for consenting FAST stages 2-3 subjects: FAST stages 2-3 participants are usually competent to make medical and legal decisions, and will be consented directly, unless there is a caregiver, legally appointed representative, or other reason to think that an informed consent cannot be given by the participants without approval by a reliable informant acting on their behalf.
* Considerations for consenting FAST stage 4 (mild dementia) participants: FAST stage 4 participants will be consented by having them give oral or written assent, indicating their preference with regard to study participation. In addition, the caregiver or legally appointed representative of a demented participants will be consented to assure full understanding of study procedures and willingness on behalf of the participants to participate in the study.

This approach has been evaluated by the Department of Psychiatry and Behavioral Sciences at Johns Hopkins, and found to adequately ensure informed consent (Black et al. 2010). They concluded that ADRD participants should not be excluded from study participation if they cannot directly consent themselves, so long as their caregivers can consent, and the participants can assent, either verbally or in writing, their preference to participate in the study.

The caregiver or legally appointed representative will be required to accompany participants to participate in the required procedures. A copy of the appropriate document (e.g., the power of attorney for healthcare) will be obtained and filed with the original ICF.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be age 50 and older (no age upper limit) at time of informed consent.
* Adults of any gender, race or ethnicity are eligible to enroll in the study.
* Participants must have cognitive impairment as demonstrated by a Memory Performance Index (MPI) of 50 or below, or delayed free recall score of 6 or below if MPI is greater than 50.
* Participants must have a FAST stage of 2-4.
* Participants with FAST Stage 4 must have the caregiver or legally appointed representative who can provide an appropriate documents (e.g., the power of attorney for healthcare)
* Participants must be proficient in spoken and written English for consenting as well as for study participation since the intervention in this study (e.g., coaching program) is currently only available in English.
* Participants with medical conditions must be stable for these conditions. Stable control on medication is acceptable.
* Participants, with or without assistance, must be able to use a computer and web interface. If assistance is needed, it must be readily available to them.
* Participants must be able to converse with a coach telephonically. Telephone coaching is part of data-driven health coaching.
* Participants must have regular access to a computer and the Internet along with dedicated email address since certain aspects of the program (e.g. cognitive training) are delivered electronically.
* Participants must have normal visual acuity (or corrected to normal) and normal color vision as indicated by self-report
* Participants must have adequate hearing acuity as indicated by self-report
* Participants must have adequate motor capacity to use a mobile device/iPad/computer as indicated by self-report

Exclusion Criteria:

* Participants with an existing diagnosis of a non-AD neurodegenerative disorder (e.g., Lewy Body Disease, Frontal-Temporal Disease).
* Participants with a diagnosis of cerebrovascular disease as the primary cause of cognitive impairment.
* Participants who have participated in the Arivale program or the HPWP. These employed coaching similar to the approach that will be used in the current study.
* A previously reported AD high-risk mutation (e.g., in the PSEN or APP genes) in the participant or immediate family (children, siblings, or parents). Such patients may accumulate amyloid faster than in late onset AD, and therefore may show less pronounced benefit from intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Coaching for Cognitive Decline | 2 years
  Test the hypothesis that coaching is better than no coaching for people in the early stages and at risk for cognitive decline. We plan to test that after two years of coaching, participants in the coaching arm will have higher cognitive scores as measured by the MCI score.
  Participants in COCOA will be assessed with the MCIS, which quantifies cognition with the Memory Performance Index (MPI) component score on a 0 to 100 scale (below normal: <50). The MPI will be our primary outcome measure for cognitive function. It is quick and inexpensive to administer. The MPI score is sensitive to slight cognitive deficits, and thus serves as an excellent single measure of cognition to serve as one of our two primary outcome measures Development and validation of the Memory Performance Index: reducing measurement error in recall tests.

SECONDARY OUTCOMES:
Diagnosis of Alzheimer's Disease | 2 years
  Measure transition from early and moderate cognitive decline into clinically diagnosed Alzheimer's disease. Our other primary outcome measure is the Functional Assessment Staging Test (FAST) to evaluate overall disease progression. FAST produces ordinal classification (7 major stages, 1-7, with 11 sub-stages, 6a to e and 7a to f. Higher ordinal numbers represent worse outcomes than lower original numbers. Within an equivalent ordinal number, later letters of the alphabet represent worse outcomes. (Sclan SG, Reisberg B. Functional assessment staging (FAST) in Alzheimer's disease: reliability, validity, and ordinality. Int. Psychogeriatr. 1992;4 Suppl 1:55-69)
Memory Performance Index | 2 years
  The Memory Performance Index is a quantitative measure of cognitive function. The MPI scale ranges from 0 to 100. It is a component of the MCI Screen. The MCI Screen's components measure the respondent's performance in terms of: pattern of words recalled immediately and after a delay attention and concentration, judgment and reasoning, and short term memory.
FAST Stage | 2 years
  The Functional Assessment Staging Test (FAST) measures functional status. FAST Stage 1 is normal. Other stages correspond to: cognitive impairment without functional impairment (FAST 2), cognitive impairment with functional impairment but without impairment in instrumental activities of daily living (FAST 3, also known as mild cognitive impairment, MCI), or cognitive impairment with impaired instrumental activities of daily living (FAST 4). Measures the effect of the intervention on functional status. FAST stage 4 is a surrogate for a clinical diagnosis of Alzheimer's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Andres, MA, Study Director — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: Undecided